CLINICAL TRIAL: NCT04487795
Title: Age-related Changes of Crystalline Lens Tilt and Decentration: A Swept-source Optical Coherence Tomography Study
Status: Completed | Type: Observational
Sponsor: Yune Zhao (Other)
Responsible Party: Sponsor-Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: SSOCT-lens tilt
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Crystalline Cataract; Lens; Anomaly
Keywords: crystalline lens tilt; crystalline lens decentration; swept-source optical coherence tomography
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- under 18 years old
- 18-40 years old
- 41-60 years old
- over 60 years old

SUMMARY:
230 participants at Eye Hospital of Wenzhou Medical University during June, 2019 and August, 2019 were enrolled in this study. 230 right eyes and 88 left eyes were included for the measurement. All the measurements were performed under non-mydriatic conditions in a dim examination room using the CASIA2 swept-source AS-OCT system.

ELIGIBILITY:
Inclusion Criteria：

* healthy volunteers and patients with age-related cataract

Exclusion Criteria:

* aphakia or pseudophakia
* any other ocular diseases with the exception of senile cataract
* any history of ocular surgery
* fixation difficulties caused by any reasons

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers and patients with age-related cataract at Eye hospital of Wenzhou Medical University
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-17 (Actual)

PRIMARY OUTCOMES:
crystalline lens tilt | 2020.4.30
  magnitude and direction of crystalline lens lilt
crystalline lens decentration | 2020.4.30
  magnitude and direction of crystalline lens decentration

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang, China